CLINICAL TRIAL: NCT01357889
Title: A Multidose Study in Subjects With Type 2 Diabetes Mellitus to Assess the Pharmacokinetics and Pharmacodynamics of Albiglutide
Brief Title: Pharmacokinetics/Pharmacodynamics of Albiglutide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114856
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacokinetics; pharmacodynamics; GSK716155; albiglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- process 2 albiglutide (Active Comparator): albiglutide 30mg from process 2 drug substance
  Interventions: Biological: albiglutide (GSK716155)
- process 3 albiglutide (Active Comparator): albiglutide 30mg from process 3 drug substance
  Interventions: Biological: albiglutide (GSK716155)

INTERVENTIONS:
Biological: albiglutide (GSK716155) — subcutaneous injection administered once a week
  Other Names: process 2
  Arms: process 2 albiglutide
Biological: albiglutide (GSK716155) — subcutaneous injection administered once a week
  Other Names: process 3
  Arms: process 3 albiglutide

SUMMARY:
The first part of the study includes a single dose treatment period to evaluate the pharmacokinetic bioequivalence of a subcutaneous injection of albiglutide from process 2 drug substance compared with process 3 drug substance. The second part of the treatment period will evaluate additional pharmacokinetic and pharmacodynamic parameters and safety and tolerability of repeat doses of albiglutide given weekly for 12 weeks from process 2 drug substance compared with process 3 drug substance. Subjects with type 2 diabetes whose glycemia is inadequately controlled on their current regimen of diet and exercise or stable dose of metformin will be recruited into the study.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter, 2 parallel group study. The first part of the treatment period will evaluate the pharmacokinetic bioequivalence of a single dose of a subcutaneous injection of 30mg of albiglutide from process 2 drug substance compared with process 3 drug substance. The second part of the treatment period will evaluate additional pharmacokinetic parameters, pharmacodynamic parameters, immunogenicity, effects on glycosylated hemoglobin and fasting plasma glucose, and safety and tolerability of repeat doses of subcutaneous injections of 30mg of albiglutide given weekly for 12 weeks from process 2 drug substance compared with process 3 drug substance. Subjects with type 2 diabetes whose glycemia is inadequately controlled on their current regimen of diet and exercise or stable dose of metformin will be recruited into the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a historical diagnosis of type 2 diabetes mellitus who are experiencing inadequate glycemic control on their current regimen of diet and exercise or on a stable dose of metformin
* Body mass index ≥20 kg/m2 and ≤45 kg/m2
* Fasting C-peptide ≥0.8 ng/mL (≥0.26 nmol/L)
* Thyroid-stimulating hormone level is normal or clinically euthyroid
* Female subjects of childbearing potential (i.e., not surgically sterile and/or not postmenopausal) must be practicing adequate contraception.

Exclusion Criteria:

* Current ongoing symptomatic biliary disease or history of pancreatitis
* History of significant GI surgery
* Recent clinically significant cardiovascular and/or cerebrovascular disease
* History of human immunodeficiency virus infection
* History of, or current hepatic disease
* History of alcohol or substance abuse
* Female subject is pregnant, lactating, or <6 weeks postpartum
* History of type 1 diabetes
* Receipt of any investigational drug within the 30 days, or 5 half-lives whichever is longer, before Screening or a history of receipt of an investigational antidiabetic drug within the 3 months before randomization, or receipt of any GLP-1 agents including albiglutide
* History of, or family history of thyroid disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (28):
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Mason, Ohio
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Lewisburg, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114856 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114856 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114856 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114856 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114856 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114856 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114856 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment number reflects the 283 participants starting the Multiple-dose Phase.
Pre-assignment Details: This study was comprised of a Screening Period (up to 2 weeks), a Run-in Period (4 weeks), a Treatment Period (TP: 17 weeks), and a Follow-up (8 weeks) Period. The TP had a Single-dose Phase (Bioequivalence [BE] Phase: 28 days) and a 12-week Multiple-dose Phase. In the BE Phase, 186 participants were randomized; 167 received >=1 treatment dose.
Groups:
- Albiglutide Process 2: During the BE Phase, participants received a single dose of albiglutide 30 milligrams (mg) from the Process 2 drug product, injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen. After completing the BE phase, participants progressed into the Multiple-dose Phase of the study, beginning at Week 5, during which participants received 12 weekly injections of albiglutide 30 mg from the Process 2 drug product, injected subcutaneously into the abdomen, alternating between the right and left sides of the body, using a fixed-dose, prefilled, single-use injector pen. Additional participants (other than those completing the BE Phase and progressing to the Multiple-dose Phase) were randomized into the Multiple-dose Phase of the study. All participants returned for the 8-week post-treatment follow-up visit.
- Albiglutide Process 3: During the BE Phase, participants received a single dose of albiglutide 30 mg from the Process 3 drug product, injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen. After completing the BE phase, participants progressed into the Multiple-dose Phase of the study, beginning at Week 5, during which participants received 12 weekly injections of albiglutide 30 mg from the Process 3 drug product, injected subcutaneously into the abdomen, alternating between the right and left sides of the body, using a fixed-dose, prefilled, single-use injector pen. Additional participants (other than those completing the BE Phase and progressing to the Multiple-dose Phase) were randomized into the Multiple-dose Phase of the study. All participants returned for the 8-week post-treatment follow-up visit.
Period: Single-dose Phase (BE Phase: 28 Days)
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Started | 86 | 81
Completed | 82 | 79
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Persistent Hyperglycemia | 1 | 1
Not completed — Physician Decision | 1 | 0
Period: Multiple-dose Phase (MDP) (Overall)
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Started | 141 (After completion of the BE Phase, additional participants were randomized to the Overall Phase.) | 142 (After completion of the BE Phase, additional participants were randomized to the Overall Phase.)
Completed | 125 | 126
Not Completed | 16 | 16
Not completed — Adverse Event | 2 | 2
Not completed — Noncompliance | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawn Due to Hyperglycemia | 7 | 7
Period: Follow-up Phase (FUP) (8 Weeks)
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Started | 141 (All participants who started the MDP entered the FUP, regardless of MDP completion status.) | 142 (All participants who started the MDP entered the FUP, regardless of MDP completion status.)
Completed | 138 | 138
Not Completed | 3 | 4
Not completed — Noncompliance | 1 | 0
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Hyperglycemia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Albiglutide Process 2: During the BE Phase, participants received a single dose of albiglutide 30 mg from the Process 2 drug product, injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen. After completing the BE phase, participants progressed into the Multiple-dose Phase of the study, beginning at Week 5, during which participants received 12 weekly injections of albiglutide 30 mg from the Process 2 drug product, injected subcutaneously into the abdomen, alternating between the right and left sides of the body, using a fixed-dose, prefilled, single-use injector pen. Additional participants (other than those completing the BE Phase and progressing to the Multiple-dose Phase) were randomized into the Multiple-dose Phase of the study. All participants returned for the 8-week post-treatment follow-up visit.
- Total: Total of all reporting groups
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3 | Total
Number analyzed (Participants) | 141 | 142 | 283
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data are reported for participants randomized to the Single- and Multiple-dose Phases (Overall).
  Years | 52.6 (11.18) | 54.4 (10.53) | 53.5 (10.88)
Gender [Count of Participants; unit: Participants] — Baseline data are reported for participants randomized to the Single- and Multiple-dose Phases (Overall).
  Participants
    Female | 78 | 76 | 154
    Male | 63 | 66 | 129
Race/Ethnicity, Customized [Number; unit: Participants] — Baseline data are reported for participants randomized to the Single- and Multiple-dose Phases (Overall).
  Participants
    African American/African Heritage | 15 | 20 | 35
    American Indian or Alaskan Native | 0 | 1 | 1
    Asian - Central/South Asian Heritage | 2 | 0 | 2
    Asian - East Asian Heritage | 1 | 2 | 3
    Asian - South East Asian Heritage | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    White - White/Caucasian/European Heritage | 120 | 117 | 237

OUTCOME MEASURES:

1. Secondary Outcome: Trough (Pre-dose) Plasma Concentrations of Albiglutide in the Mutiple-dose Phase (MDP)
Description: The trough concentration of albiglutide at Week 5, Week 9, Week 13, Week 17 (EOT), and Week 25 (Follow-up) following multiple-dose administration was estimated. The time and date of sample collection pre-dose was to be recorded.
Time Frame: Immediately pre-dose at Week 5, Week 9, Week 13, Week 17 (End of Treatment [EOT]), and Week 25 (Follow-up)
Population: PK Concentration Population (PKCP): participants (par.) in the MDP for whom a PK sample was collected/analyzed. Only par. available at the specified time points were analyzed (n= X, X in the category titles). Different par. may have been analyzed at different time points; the overall number of par. analyzed reflects everyone in the PKCP.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 136 | 138
ng/mL
  Week 5, n=131, 135 | 10.55 (34.847) | 8.70 (25.547)
  Week 9, n=127, 130 | 2420.95 (1064.204) | 2519.62 (911.794)
  Week 13, n=126, 127 | 2352.94 (984.488) | 2356.27 (987.143)
  Week 17 (EOT), n=123, 125 | 2360.19 (1005.598) | 2436.63 (1089.381)
  Week 25 (follow-up), n=121, 123 | 28.20 (291.287) | 14.45 (160.245)

2. Secondary Outcome: Number of Participants With Anti-albiglutide Antibody Formation at Baseline and Weeks 5, 9, 13, 17, and 25 in the Multiple-dose Phase
Description: The presence of anti-albiglutide antibodies after repeat-dose administration was assessed using a qualified enzyme-linked immunosorbent assay. The assay involved screening, confirmation, and titration steps (tiered-testing approach). The number of participants who tested positive for anti-albiglutide antibodies are presented by visit.
Time Frame: Baseline, Week 5, Week 9, Week 13, Week 17, and Week 25 (Follow-up)
Population: Safety Population: all par. who received at least 1 dose of study medication. Only those par. available at the specified time points were analyzed (represented by n= X, X in the category titles). Different par. may have been analyzed at different time points, so the overall number of par. analyzed reflects everyone in the Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 141 | 142
Participants
  Baseline, n=139, 140 | 1 | 0
  Week 5, n=131, 132 | 1 | 0
  Week 9, n=124, 120 | 0 | 0
  Week 13, n=119, 122 | 1 | 3
  Week 17, n=119, 127 | 0 | 5
  Week 25, n=116, 118 | 0 | 2

3. Secondary Outcome: AUC (0-last) and AUC (0-inf) of Albiglutide in the BE Phase
Description: The area under the concentration-time (AUC) curve from time zero to the last quantifiable concentration (0-last) and AUC (0-inf) of albiglutide in the BE Phase were measured. AUC is a measure of how much albiglutide is in the blood at certain time points. Blood samples for PK analysis were collected prior to dosing at Baseline and 24 hr, 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hr, 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: Albiglutide PK Population. Participants with insufficient concentration data or an unestimable terminal elimination rate constant were excluded from analysis. Different par. may have been analyzed at different time points; the overall number of par. analyzed reflects everyone in the PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter
Groups:
- Albiglutide Process 2: During the BE Phase, participants received a single dose of albiglutide 30 milligrams (mg) from the Process 2 drug product, injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen.
- Albiglutide Process 3: During the BE Phase, participants received a single dose of albiglutide 30 mg from the Process 3 drug product, injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen.
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 85 | 80
nanograms*hour/milliliter
  AUC (0-last), n=84, 80 | 447294.0 (55.5) | 426263.5 (45.2)
  AUC (0-inf), n=75, 74 | 496190.2 (41.8) | 464985.4 (39.7)

4. Secondary Outcome: Tmax and Tlag of Albiglutide in the BE Phase
Description: Time of the maximum observed plasma concentration (tmax) and the observed time prior to the first quantifiable plasma concentration (tlag) of albiglutide in the BE Phase were measured. Blood samples for PK analysis were collected prior to dosing at Baseline and 24 hr, 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hr, 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: Albiglutide PK Population. Participants with insufficient concentration data or terminal elimination rate constant not estimable were excluded.
Measure: Median (Full Range); unit: Hours
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 85 | 80
Hours
  tmax, n=85, 80 | 95.50 [23.4 to 214.3] | 96.08 [20.5 to 217.8]
  tlag, n=84, 80 | 0.00 [0.0 to 24.1] | 0.00 [0.0 to 24.1]

5. Secondary Outcome: Cmax of Albiglutide in the BE Phase
Description: Cmax of albiglutide in the BE Phase was measured. Blood samples for PK analysis were collected prior to dosing at Baseline and 24 hr, 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hr, 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: Albiglutide PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 85 | 80
ng/mL | 1881.05 (58.3) | 1743.05 (49.1)

6. Secondary Outcome: t1/2 of Albiglutide in the BE Phase
Description: The terminal elimination half-life (t1/2) of albiglutide in the BE Phase was measured. Blood samples for PK analysis were collected prior to dosing at Baseline and 24 hr, 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hr, 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: Albiglutide PK Population. Participants with insufficient concentration data or an unestimable terminal elimination rate constant were excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 75 | 74
Hours | 106.42 (16.3) | 113.83 (22.5)

7. Secondary Outcome: Apparent Clearance of Albiglutide in the BE Phase
Description: The apparent clearance (CL/F) of albiglutide in the BE Phase was measured. Blood samples for PK analysis were collected prior to dosing at Baseline and 24 hr, 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hr, 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 75 | 74
Liters per hour | 0.06046 (41.8) | 0.06452 (39.7)

8. Secondary Outcome: Apparent Volume of Distribution in the Terminal Phase of Albiglutide in BE Phase
Description: The apparent volume of distribution in the terminal phase (V/F) of albiglutide in the BE Phase was measured. Blood samples for PK analysis were collected prior to dosing at Baseline and 24 hr, 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hr, 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 75 | 74
Liters | 9.283 (44.0) | 10.595 (44.3)

9. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 17
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. This analysis used the last observation carried forward (LOCF) method for missing post-Baseline HbA1c values. HbA1c values obtained after hyperglycemic rescue were treated as missing and replaced with pre-rescue values. Baseline is defined as the last available assessment on or prior to the day on which the first dose of study drug was received. Based on analysis of covariance (ANCOVA): Change = treatment + Baseline HbA1c + age category + weight category + background antidiabetic therapy category.
Time Frame: Baseline and Week 17
Population: Efficacy Population - LOCF: all participants who received a dose of study medication and who had a Baseline measurement and at least 1 post-Baseline HbA1c or fasting plasma glucose (FPG) measurement. Only participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in blood
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 135 | 135
Percentage of HbA1c in blood | -0.75 (0.082) | -0.84 (0.082)

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 17
Description: This analysis used the LOCF method for missing post-Baseline FPG values. FPG values obtained after hyperglycemic rescue were treated as missing and replaced with pre-rescue values. Baseline is defined as the last available assessment on or prior to the day on which the first dose of study drug was received. Based on ANCOVA: Change = treatment + Baseline FPG + age category + weight category + background antidiabetic therapy category.
Time Frame: Baseline and Week 17
Population: Efficacy Population - LOCF
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 141 | 141
millimoles per liter | -1.11 (0.231) | -1.21 (0.231)

11. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs. Hypoglycemic events are excluded from this table, except for serious adverse events.
Time Frame: From the time the participant consented to participate in the study through Visit 28 (Week 25) or the final follow-up visit, for participants who discontinued active participation in the study
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 141 | 142
Participants
  Any AE | 106 | 91
  Any SAE | 5 | 1

12. Secondary Outcome: Number of Participants With Indicated Adverse Events of Special Interest
Description: Adverse events of special interest included cardiovascular events, hypoglycemic events, pancreatitis events, thyroid events, gastrointestinal (GI) events, diabetic retinopathy events, systemic allergic reactions (SAR), injection site reactions (ISR), and liver events (AEs from investigations and hepatobiliary disorders were considered).
Time Frame: From the time the participant consented to participate in the study through Visit 28 (Week 25) or the final follow-up visit, for participants who discontinue active participation in the study
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 141 | 142
Participants
  Any cardiovascular AE | 15 | 9
  Any hypoglycemic AE | 11 | 7
  Any thyroid AE | 2 | 1
  Any GI AE | 36 | 32
  Any SAR AE | 1 | 0
  Any ISR AE | 13 | 7
  Any hepatobiliary AE | 2 | 2
  Any investigations | 5 | 10
  Any pancreatitis AE | 0 | 0
  Any diabetic retinopathy AE | 0 | 0

13. Secondary Outcome: Number of Participants With a Change From Baseline of Clinical Concern in Hematology Values by Any On-therapy Visit
Description: Criteria for values of potential concern were determined by the medical monitors. For hematocrit, a >0.1 decrease from Baseline was considered to be of clinical concern. For hemoglobin, a >25 grams per liter (g/L) decrease from Baseline was considered to be of clinical concern.
Time Frame: Week 1 through Week 25
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 140 | 140
Participants
  Hematocrit >0.1 decrease | 1 | 0
  Hemoglobin >25 g/L | 1 | 1

14. Secondary Outcome: Number of Participants With a Change From Baseline of Clinical Concern in Vital Signs by Any On-therapy Visit
Description: Vital signs measured included systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. Criteria for values of potential concern were determined by the medical monitors. For SBP, a decrease or increase >30 millimeters of mercury (mmHg) from Baseline was considered to be of clinical concern. For DBP, a decrease or increase >20 mmHg from Baseline was considered to be of clinical concern. For heart rate, a decrease or increase >30 beats per minute (bpm) was considered to be of clinical concern.
Time Frame: Week 1 through Week 25
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 141 | 141
Participants
  SBP, decrease >30 mmHg | 18 | 16
  SBP, increase >30 mmHg | 10 | 10
  DBP, decrease >20 mmHg | 19 | 16
  DBP, increase >20 mmHg | 7 | 8
  Heart rate, decrease >30 bpm | 1 | 4
  Heart rate, increase >30 bpm | 5 | 4

15. Secondary Outcome: Number of Participants With the Indicated Change From the Screening Assessment in Physical Examination at Week 17
Description: A complete physical examination was performed at Screening and at Week 17 and included evaluation of the following organ or body systems: skin (including injection site); head; eyes; ears, sose, and throat (ENT); thyroid; respiratory system; cardiovascular system; abdomen (liver, spleen); lymph nodes; central nervous system (CNT); and extremities. The assessment was categorized as improved, no change, worsened, and not done.
Time Frame: Screening and Week 17
Population: Safety Population. Only participants analyzed at Week 17 are presented.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 120 | 125
Participants
  Skin, Improved | 2 | 3
  Skin, No Change | 112 | 117
  Skin, Worsened | 6 | 4
  Skin, Not done | 0 | 1
  Head, Eyes, ENT, Improved | 3 | 0
  Head, Eyes, ENT, No Change | 115 | 122
  Head, Eyes, ENT, Worsened | 2 | 2
  Head, Eyes, ENT, Not done | 0 | 1
  Cardiovascular system, Improved | 1 | 0
  Cardiovascular system, No Change | 119 | 124
  Cardiovascular system, Worsened | 0 | 0
  Cardiovascular system, Not done | 0 | 1
  Respiratory system, Improved | 0 | 1
  Respiratory system, No Change | 120 | 123
  Respiratory system, Worsened | 0 | 0
  Respiratory system, Not done | 0 | 1
  Abdomen (Liver and Spleen), Improved | 0 | 0
  Abdomen (Liver and Spleen), No Change | 120 | 121
  Abdomen (Liver and Spleen), Worsened | 0 | 3
  Abdomen (Liver and Spleen), Not done | 0 | 1
  Lymph Nodes, Improved | 0 | 0
  Lymph Nodes, No Change | 120 | 123
  Lymph Nodes, Worsened | 0 | 0
  Lymph Nodes, Not done | 0 | 2
  CNS, Improved | 1 | 2
  CNS, No Change | 118 | 122
  CNS, Worsened | 1 | 0
  CNS, Not done | 0 | 1
  Extremities, Improved | 4 | 1
  Extremities, No Change | 114 | 118
  Extremities, Worsened | 2 | 4
  Extremities, Not done | 0 | 2
  Thyroid, Improved | 0 | 0
  Thyroid, No Change | 120 | 123
  Thyroid, Worsened | 0 | 0
  Thyroid, Not done | 0 | 2

16. Secondary Outcome: Number of Participants With a Change From Baseline of Clinical Concern in Electrocardiogram (ECG) Values by Any On-therapy Visit
Description: ECG parameters include heart rate, QRS interval, QTinterval, QT interval - Bazett correction (QTcB), QT interval - Fridericia correction (QTcF), RR interval, and PR interval. Criteria for values of potential concern were determined by the medical monitors. For the QRS interval, an increase of >25% when Baseline QRS >100 milliseconds (msec) and an increase of >50% when Baseline QRS <=100 msec was considered to be of clinical concern. For QTcF, a >=60 msec change from Baseline was considered to be of clinical concern. For the PR interval, an increase of >25% when Baseline PR >200 msec and an increase of >50% when Baseline PR <=200 msec was considered to be of clinical concern.
Time Frame: Week 1 through Week 25
Population: Safety Population. Only those participants available at the specified time points were analyzed. Different par. may have been analyzed at different time points; the overall number of par. analyzed reflects everyone in the Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 141 | 142
Participants
  QRS, Increase of > 25% or >50%, n=139, 137 | 1 | 0
  QTcF, >=60 msec, n=139, 137 | 0 | 0
  PR, Increase of > 25% or >50%, n=137, 135 | 0 | 0

17. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time Zero to Infinity (0-inf) of Albiglutide in the Bioequivalence (BE) Phase
Description: To assess the bioequivalence of the two formulations of albiglutide, an analysis of variance (ANOVA) model with treatment as a fixed effect was applied to the natural-log-transformed parameter AUC(0-inf) estimated from the BE Phase. AUC is a measure of how much albiglutide is in the blood at certain time points. The Process 2 treatment group (albiglutide derived from process 2) was the reference group and was compared with the Process 3 treatment group (albiglutide derived from process 3) as the test group (i.e., treatment comparisons based on the ratio of Process 3:Process 2). Blood samples for pharmacokinetic analysis were collected prior to dosing at Baseline and 24 hours (hr), 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hours (hr), 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: Albiglutide Pharmacokinetic (PK) Population: all participants who had sufficient samples to calculate PK parameters of albiglutide. Participants with insufficient concentration data or an unestimable terminal elimination rate constant were excluded from analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 75 | 74
nanograms*hour/milliliter | 496190.200 (42) | 464985.355 (40)
Statistical Analysis 1: Comparison: Albiglutide Process 2 vs Albiglutide Process 3; Test type: Non-Inferiority or Equivalence — To establish BE, the 90% CI for the ratio of Process 3 (P3) to Process 2 (P2) geometric least squares means (LSMs) for AUC (0-inf) must have fallen within the BE limit of 0.8 and 1.25; ANOVA; Ratio of Geometric LSMs (P3:P2) = 0.937, 90% CI 2-sided [0.842 to 1.042]

18. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Albiglutide in the BE Phase
Description: To assess the bioequivalence of the two formulations of study drug, an analysis of variance (ANOVA) model with treatment as a fixed effect was applied to the natural-log-transformed parameter Cmax estimated from the BE phase. The Process 2 treatment group (albiglutide derived from process 2) was the reference group and was compared with the Process 3 treatment group (albiglutide derived from process 3) as the test group (i.e., treatment comparisons based on the ratio of Process 3:Process 2). Blood samples for pharmacokinetic analysis were collected prior to dosing at Baseline and 24 hours (hr), 48 hr, 96 hr, 120 hr, 216 hr, 312 hr, 480 hr, and 672 hr after administration of the Baseline study medication.
Time Frame: Pre-dose at Baseline; 24 hr, 48 hr, 96 hr, 216 hr, 312 hr, 480 hr, and 672 hr post-dose
Population: Albiglutide PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Number analyzed (Participants) | 85 | 80
nanograms per milliliter (ng/mL) | 1881.053 (58) | 1743.053 (49)
Statistical Analysis 1: Comparison: Albiglutide Process 2 vs Albiglutide Process 3; Test type: Non-Inferiority or Equivalence — To establish BE, the 90% CI for the ratio of Process 3:Process 2 geometric least squares means for Cmax must have fallen within the BE limit of 0.8 and 1.25; ANOVA; Ratio of Geometric LSMs (P3:P2) = 0.927, 90% CI 2-sided [0.813 to 1.056]

ADVERSE EVENTS:
Time Frame: On-therapy SAEs/non-serious AEs (onset on/after study drug start date and within 56 days after last dose) were collected from time of study participation consent through Week 25/final follow-up visit for par. who discontinued active study participation.
Description: SAEs and non-serious AEs are reported for members of the Single- and Multiple-dose Phases Safety Population, comprised of all participants who received at least 1 dose of study medication.
Arm/Group | Albiglutide Process 2 | Albiglutide Process 3
Serious Adverse Events (participants affected / at risk) | 5/141 | 1/142
Other Adverse Events (participants affected / at risk) | 84/141 | 69/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide Process 2 (N=141) | Albiglutide Process 3 (N=142)
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide Process 2 (N=141) | Albiglutide Process 3 (N=142)
Upper respiratory tract infection (Infections and infestations) | 6 | 8
Nasopharyngitis (Infections and infestations) | 15 | 4
Sinusitis (Infections and infestations) | 9 | 4
Urinary tract infection (Infections and infestations) | 5 | 4
Gastroenteritis viral (Infections and infestations) | 6 | 3
Otitis media (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 6 | 2
Nausea (Gastrointestinal disorders) | 11 | 13
Diarrhoea (Gastrointestinal disorders) | 11 | 8
Vomiting (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Flatulence (Gastrointestinal disorders) | 0 | 4
Gastooesophageal reflexu disease (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 4 | 4
Injection site haematoma (General disorders) | 1 | 4
Chest pain (General disorders) | 1 | 3
Injection site reaction (General disorders) | 8 | 2
Injection site rash (General disorders) | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 6
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 6
Headache (Nervous system disorders) | 13 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Hypertension (Vascular disorders) | 4 | 5
Palpitations (Cardiac disorders) | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Lipase increased (Investigations) | 1 | 4
Amylase increased (Investigations) | 0 | 4
Seasonal allergy (Immune system disorders) | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.